CLINICAL TRIAL: NCT00972686
Title: A Phase I Open-Label, Dose-Escalation Study of the Phosphoinositide 3-Kinase Inhibitor GSK2126458 in Subjects With Solid Tumors or Lymphoma
Brief Title: Dose-Escalation Study of GSK2126458
Acronym: FTIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112826
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Solid Tumours
Keywords: solid tumors; lymphoma; Phosphoinositide 3-kinase inhibitor
MeSH Terms: conditions — Lymphoma | interventions — omipalisib

ARMS (1):
- GSK2126458 (Experimental): GSK2126458 will be dosed continuously (every day) for the duration a 28 day cycle. The 28 day cycles will continue until the subjects withdraw from the study.
  Interventions: Drug: GSK2126458

INTERVENTIONS:
Drug: GSK2126458 — GSK2126458 is an experimental treatment for patients with cancer.

SUMMARY:
P3K112826 is a Phase I, first-time-in-human dose escalation study in subjects with refractory malignancy. The primary objective of this study is to determine the recommended Phase II dose of GSK2126458 based on safety and tolerability, pharmacokinetics, pharmacodynamics and preliminary evidence of clinical activity. Secondary objectives are to characterize the pharmacokinetics of GSK2126458; and to explore relationships between GSK2126458 pharmacokinetics, pharmacodynamics, response prediction biomarkers and clinical endpoints.

DETAILED DESCRIPTION:
This study is a Phase I, first-time-in-human dose escalation study in subjects with refractory solid tumors or lymphoma. The primary objective of this study is to determine the recommended Phase II dose of GSK2126458 based on safety and tolerability, pharmacokinetics, pharmacodynamics and preliminary evidence of clinical activity. Secondary objectives are to characterize the pharmacokinetics of GSK2126458; and to explore relationships between GSK2126458 pharmacokinetics, pharmacodynamics, response prediction biomarkers and clinical endpoints.

Subjects with solid tumors or lymphoma will initially receive oral GSK2126458 daily for 28 consecutive days in each 28 day cycle. Subjects may be dosed once or twice a day or may be dosed on an intermittent schedule depending on the safety, pharmacokinetic and pharmacodynamic results that become available as the study progresses. The starting dose will be 0.1 mg once a day. Expansion of some cohorts will be conducted to test tumor pharmacodynamics, further explore the toxicity profile and to look for preliminary evidence of activity in subjects with tumors with PIK3CA mutations. The recommended Phase II dose will be the lowest dose explored (at or below MTD) that maintains biologic activity with an acceptable tolerability profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed diagnosis of solid tumor malignancy, or lymphoma
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Female or male that is willing to take measures to avoid pregnancy in self or a partner, including abstinence, or double barrier method.
* Adequate organ system function

Exclusion Criteria:

* Use of an investigational anti-cancer medication within 28 days or 5 half-lives preceding the first dose of GSK2126458.
* Chemotherapy within the last 3 weeks (6 weeks for prior nitrosourea or mitomycin C
* Any major surgery, radiotherapy, or immunotherapy within the last 4 weeks.
* Prior use of any PI3K inhibitor.
* Current use of a prohibited medication or requires any of these medications during treatment with GSK2126458.
* Presence of an active gastrointestinal disease or other condition known to interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* Unresolved toxicity greater than Grade 1 from previous anti-cancer therapy except alopecia.
* QTc interval ≥ 480 msecs.
* History of acute coronary syndromes; Class II, III, or IV heart failure; stroke or subarachnoid hemorrhage.
* Systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg.
* Previously diagnosed Type 1 diabetes mellitus. Subjects with Type 2 diabetes are prohibited in the dose escalation part of the study.
* Symptomatic or untreated leptomeningeal or brain metastases.
* Primary malignancy of the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2012-12-12 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and changes in laboratory values and vital signs. Pharmacokinetic parameter values for GSK2126458, Change from baseline in protein markers in tumor and/or blood. Blood glucose and insulin levels. Tumor response, RECIST defined | Subjects continue on study until disease progression or consent withdrawal

SECONDARY OUTCOMES:
Metabolic profile in plasma at the maximum tolerated dose | Subjects continue on study until disease progression or consent withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (7):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112826 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112826?search=study&b'search_terms=112826'#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112826 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register